CLINICAL TRIAL: NCT01521052
Title: Evaluation of the H-Coil Transcranial Magnetic Stimulation (TMS) Device - Safety and Feasibility Study for Treatment of Major Depressive Episode in the Elderly
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHA-0001-11
Record Dates: First submitted 2012-01-25; First posted 2012-01-30 (Estimated); Last update posted 2012-01-30 (Estimated); Status verified 2012-01

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- elderly depressed patients (Experimental): Twenty seven (27) patients aged 68 years or above, currently suffering from a major depressive episode, who did not respond to treatment with at least one antidepressant medications in the recommended dosage and duration, or could not tolerate at least two antidepressants.
  Interventions: Device: dTMS treatment (H1 Coil)

INTERVENTIONS:
Device: dTMS treatment (H1 Coil) — All subjects will receive prefrontal deep rTMS of H1 Coil (42 trains of 2 seconds, 10 Hz, with 20 seconds inter-train intervals, up to 120% of motor threshold), for 4 weeks, 5 days a week, overall 20 sessions.

SUMMARY:
Purpose: To evaluate the safety and anti-depressive response of the H1 Coil TMS Device in elderly patients suffering from major depressive episode.

Twenty-seven (27) treatment resistance depressed-patients, 68 years of age and above, currently in a depressive episode.All subjects will receive prefrontal deep rTMS of H1 Coil (42 trains of 2 seconds, 10 Hz, with 20 seconds inter-train intervals, up to 120% of motor threshold), for 4 weeks, 5 days a week, overall 20 sessions.Safety and efficacy tests will be conducted before starting the trial (screening), once a week for the trial duration and one month following end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed by a senior psychiatrist as suffering from major depression episode according to DSM-IV (either as a part of a unipolar or a bipolar disorder).
* Rating on HDRS ≥ 20.
* Age: 68 years and above
* Treated for the current depressive episode, at least 6 weeks per antidepressant with one antidepressant in accepted dose, without improvement, and/or intolerance to 2 antidepressants, according to medical chart and ATHF (antidepressant treatment history form) instruction guidelines.
* Gave informed consent for participation in the study.
* Negative answers on safety screening questionnaire for TMS.
* If referred by a treating psychiatrist, he or she approves of the subject's participation in the study.

Exclusion Criteria:

* Axis 2 diagnosis, which is considered prominent to the current depressive episode.
* Substantial suicidal risk as judged by the treating psychiatrist or by an independent psychiatrist.
* Attempted suicide in the past year.
* Cognitive impermanent - if MMSE < 24, patient will be further assessed , and may be excluded according to the primary investigator's discretion
* History of seizure.
* History of epilepsy or seizure in first degree relatives.
* Any CNS disorder that may increase risk of seizure significantly
* History of a significant head injury.
* History of any metal in the head (outside the mouth).
* Known history of any metallic particles in the eye, implanted cardiac pacemaker or any intracardiac lines, implanted neurostimulators, surgical clips or any medical pumps.
* History of frequent or severe headaches.
* Use of hearing aids for hearing loss.
* Known history of cochlear implants.
* History of drug abuse or alcoholism.
* Serious and unstable medical condition, which is likely to exacerbate or endanger the patient during the treatment period.
* Inadequate communication with the patient.
* Under custodial care.
* Participation in current clinical study or clinical study within 30 days prior to this study.
* Patients suffering from bipolar disorder, not currently treated by mood stabilizers
* Patients declared as legally incompetent, with an appointed physical guardian and/or cannot sign informed consent due to cognitive incompetence.

Min Age: 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Safety of the H1-Coil | One Month
  maintaining subject's pre treatment, physical and neurological status.
Clinical antidepressant response | One Month
  a decline in Hamilton depression rating scale (HDRS) from the baseline rating by 50%.

SECONDARY OUTCOMES:
Clinical antidepressant remission | One Month
  exit Hamilton Depression Rating Scale <9.
Symptomatic improvement at the end point. | One Month
  Change in Hamilton Anxiety Rating Scale (HARS), Quick Inventory of Depression Symptomatology - Self Report (QIDS-SR), Clinical Global Impression (CGI).

CONTACTS AND LOCATIONS:
Locations (1):
- Shalvata Mental Health Center, Hod HaSharon, Israel